CLINICAL TRIAL: NCT02200419
Title: Blood Conservation in Cardiac Surgery Using a Novel Transfusion Algorithm Based on Point-of-care Testing-A Stepped-wedge Cluster Randomized Controlled Trial
Brief Title: POC - Transfusion Algorithm Cardiac Study
Acronym: TACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Research Manager, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-7495-A
Record Dates: First submitted 2014-06-20; First posted 2014-07-25 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Heart Diseases
Keywords: Rotem; Point of care coagulation tests; Cardiac surgery; Vascular surgery; Cardiopulmonary bypass; Blood products; Transfusion; Viscoelastic coagulation
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transfusion Algorithm (Other): Hospitals will be randomized to the intervention arm of the study in a stratified manner.
  Interventions: Other: POC-based transfusion algorithm

INTERVENTIONS:
Other: POC-based transfusion algorithm — A transfusion algorithm based on point-of-care coagulation testing.

SUMMARY:
This multi-centre study will provide sound, generalizable data on the effectiveness of a POC-based algorithm to determine to what extent this guideline can reduce blood product transfusions. Investigators will study outcomes in 7000 patients undergoing heart surgery at 10 participating hospitals. The proposed trial addresses several important research and clinical issues and has the potential to markedly improve the transfusion management and surgical care in general of cardiac surgery patients.

The intervention will be a novel POC-based algorithm that has been shown in a pilot study by us to be associated with a substantial reduction in blood product transfusions. The algorithm will employ viscoelastic and aggregometric POC-tests and an objective measure of blood loss. The primary outcome will be avoidance of red blood cell transfusion during hospitalization. The study has a 90% power to detect a 12% increase in avoidance rate. Secondary outcomes will include avoidance of red blood cell use and other blood products (plasma, platelets, and cryoprecipitate), units of blood products transfused, and adverse clinical outcomes related to transfusion (acute kidney injury, infections, and death). Data will also be collected for future health-economics analyses.

Largely due to the limitations of existing evidence, however, such algorithms are rarely used in clinical practice. The proposed trial will provide sound, generalizable data on the effectiveness of a POC-based algorithm to guide their future use. An integrated blood management algorithm that employs POC coagulation tests will reduce blood product transfusions in cardiac surgery, thereby improving clinical outcomes.

Does an integrated blood transfusion algorithm that employs POC coagulation tests applied across a network of hospitals reduce blood transfusions and associated adverse outcomes in cardiac surgery?

DETAILED DESCRIPTION:
Despite major advances in cardiac surgery, coagulopathy continues to carry a heavy burden in cases that require the use of cardiopulmonary bypass (CPB), occurring frequently and resulting in excessive blood loss, blood product transfusions, and adverse clinical outcomes. Current management of coagulopathy is hampered by the inability of conventional laboratory tests to delineate its etiology in a timely manner, thereby precluding timely and targeted transfusion therapy. With the advent of point-of-care (POC) coagulation tests that can rapidly identify the etiology of coagulopathy, it may now be possible to reduce the burden of coagulopathy and thereby reduce transfusions and adverse outcomes. Several single-centre studies (including one by the investigator group) have found that the use of POC-based algorithms in cardiac surgery can markedly reduce blood product transfusions and by that means reduce morbidities and mortality.

ELIGIBILITY:
Hospital Inclusion:

* Participating hospitals must not currently be using a POC-based blood conservation algorithm; must have an in-hospital RBC transfusion rate of > 35% and platelet or plasma transfusion rates of > 20%; must conduct > 600 cardiac surgeries employing CPB per year; and must have commitments from departments of Anesthesia, Cardiac Surgery, and Laboratory Medicine to support the study and to abide by the algorithm
* Blood transfusion algorithm instituted as standard-of-care at participating hospitals
* All adult (≥ 18 years) patients undergoing cardiac surgery with cardiopulmonary bypass (CPB) will be included in the analysis.

Exclusion Criteria: Hospitals not meeting inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7402 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Point Of Care (POC) Transfusion Algorithm Cardiac Study | 2.5 years
  The primary outcome measure will be the proportion of patients who receive any allogeneic red blood cell (RBC) transfusion from admission before surgery to end of follow-up.

SECONDARY OUTCOMES:
Transfusion | 7 days
  Allogeneic blood products (platelets, plasma, cryoprecipitate) or coagulation factors (e.g., fibrinogen concentrate, factor VIIa), or undergo re-exploration; units of blood products transfused, nadir hemoglobin concentration (to identify changes in transfusion practice that may be unrelated to treatment of coagulopathy)
Blood loss | 24 hours
  Chest-tube drainage at 6 and 24 hours after surgery
Ventilation and hospital stay | 24 hours to 7 days
  Duration of mechanical ventilation and length of stay in the ICU and hospital
Kidney injury | 48 hours
  Incidence of acute kidney injury, defined as a ≥ 2-fold in increase in creatinine or new renal replacement therapy within 48 hours after surgery
Post operative complications | 7 days
  Arrhythmias, sternal infection, myocardial infarction, stroke, thromboembolic events, and death

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD, Principal Investigator — University Health Network, Toronto
Locations (12):
- Canada (12):
  - Dr. Charles McAdams, Calgary, Alberta
  - Blaine Achen, Edmonton, Alberta
  - Dr. Terry Waters, Vancouver, British Columbia
  - Dr. Sukhpal Brar, Vancouver, British Columbia
  - Dr. H. Grocott, Winnipeg, Manitoba
  - Dr. Summer Syed, Hamilton, Ontario
  - Dr. Christopher Harle, London, Ontario
  - Dr. Daniel Kim, Newmarket, Ontario
  - Dr. D. Tran, Ottawa, Ontario
  - Dr. F. Moussa, Toronto, Ontario
  - Dr. E. Medicis, Fleurimont, Quebec
  - Dr. J. Bussieres, Sainte-Foy, Quebec

REFERENCES:
- [Derived] Karkouti K, Callum J, Wijeysundera DN, Rao V, Crowther M, Grocott HP, Pinto R, Scales DC; TACS Investigators. Point-of-Care Hemostatic Testing in Cardiac Surgery: A Stepped-Wedge Clustered Randomized Controlled Trial. Circulation. 2016 Oct 18;134(16):1152-1162. doi: 10.1161/CIRCULATIONAHA.116.023956. Epub 2016 Sep 21. PMID 27654344